CLINICAL TRIAL: NCT06045130
Title: Characteristics of PUFAs Composition in Preterm Infants and Its Impact on Disease Prognosis
Brief Title: PUFAs in Preterm Infants
Acronym: PIPI
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-HS-050
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Necrotizing Enterocolitis; Intraventricular Hemorrhage; BPD - Bronchopulmonary Dysplasia; Sepsis; Periventricular Leukomalacia; Patent Ductus Arteriosus
Keywords: PUFAs
MeSH Terms: conditions — Enterocolitis, Necrotizing; Bronchopulmonary Dysplasia; Sepsis; Leukomalacia, Periventricular; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research endeavors to examine the critical composition of Polyunsaturated Fatty Acids (PUFAs) in premature infants across different gestational stages and under varying disease conditions, and delineate the metabolic attributes of PUFAs in premature infants and their interplay with the onset of diseases. This study anticipates furnishing a theoretical foundation for the rationalization of PUFAs supplementation in premature infants and for informing strategies related to disease prevention and management.

ELIGIBILITY:
Inclusion Criteria:

Infants born between 24 and 36 weeks of gestational age who are admitted within 24 hours of birth, including both premature and full-term newborns.

-

Exclusion Criteria:

Infants with severe congenital developmental abnormalities, those requiring external supplementation of PUFAs in addition to standard intravenous nutrition and breastfeeding, and those with a severe prognosis indicating non-survival during their hospitalization.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates born within 24 hours who were admitted to the Neonatology Department of the First Hospital of Jilin University, including premature infants born between 24 and 36 weeks of gestational age and full-term infants from September 2023 to August 2026, n
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-21 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mortality and severe complications of premature infants | before discharge
  incidence of death，NEC，PDA，BPD，IVH，PVL and sepsis

SECONDARY OUTCOMES:
Mortality | before discharge
  death
NEC | before discharge
  Bell stage II or III
PDA | before discharge
  confirmed by echocardiography
BPD | before discharge
  nasal CPAP/NIPPV or invasive ventilation requirement at 36 weeks postmenstrual age or at discharge, transfer or death if before 36 weeks
IVH | before discharge
  Papile grades 3-4
PVL | before discharge
  periventricular cysts on cranial ultrasound or magnetic resonance imaging
sepsis | before discharge
  blood culture positive